CLINICAL TRIAL: NCT01829828
Title: To Evaluate the Effectiveness of a Patient Self-reported Pain Scoring Tool and a Satisfaction Survey on Cancer Pain Management; Multicenter, Cross-sectional Study
Brief Title: The Effectiveness of a Patient Self-reported Pain Scoring Tool and a Satisfaction Survey on Cancer Pain Management
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR100835; FENPAI4097 (Other: Janssen Korea, Ltd., Korea); FEN-KOR-9052 (Other: Janssen Korea, Ltd., Korea)
Record Dates: First submitted 2013-04-08; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Pain
Keywords: Pain; Cancer pain; Self-reported pain scoring tool; Opioid analgesics
MeSH Terms: conditions — Pain; Cancer Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Inpatients with cancer pain: Inpatients admitted for cancer pain management
  Interventions: Behavioral: No intervention

INTERVENTIONS:
Behavioral: No intervention — This is an observational study with no investigational drug administered.

SUMMARY:
The purpose of this survey is to investigate the usefulness of a patient self-reported scoring tool on patient satisfaction improvement.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have no experience with the study self-reported pain scoring tool
* Patients who are able to understand and answer the pain scoring tool questions
* Patients admitted to a hospital for more than 5 days due to cancer pain
* Patients for whom their pain managing physicians completed the medical staff's survey

Exclusion Criteria:

* Patients who cannot answer the questions due to cognitive impairments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients admitted for cancer pain management
Sampling Method: Non-Probability Sample
Enrollment: 587 (Actual)
Dates: Start 2012-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Patient satisfaction with the control of cancer-related pain | At baseline
  Patients will answer on a 7-point scale how satisfied they feel about their cancer pain treatment. The scale scores range from 1 (not at all satisfied) to 7 (very much satisfied).

SECONDARY OUTCOMES:
Patient perception of pain | At baseline
  Patients will answer on an 11-point scale how much pain they feel. The scales scores range from 0 (no pain at all) to 10 (pain as bad as you can imagine).
Patient pain assessment by medical staff | At baseline
  The patient's physician will mark on an 11-point scale the intensity of the patient pain. The scale scores range from 0 (no pain at all) to 10 (pain as bad as you can imagine).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea